CLINICAL TRIAL: NCT00922077
Title: Individualized Neurodevelopmental Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Society for Disabled Children (Other)
Responsible Party: Gait Laboratory ELEPAP THESSALONIKI
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 001-Nikodelis
Record Dates: First submitted 2009-06-01; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: standard physical therapy program with emphasis on dynamic balance exercises

SUMMARY:
The purpose of the study was to evaluate this therapeutic intervention by expressing functional level with valid quantitative data.

DETAILED DESCRIPTION:
The intervention lasted 6 weeks. There were 3 sessions per week. At each session there was a part of standard physical therapy program and there was also a part with emphasis on dynamic balance exercises.

ELIGIBILITY:
Inclusion Criteria:

* spastic tetraplegia

Exclusion Criteria:

* vision problems

Ages: 6 Years to 9 Years | Sex: Female
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Society for Disabled Children, Thessaloniki, THessaloniki, Greece